CLINICAL TRIAL: NCT07114549
Title: External Validation of the MASCAN Score for the Classification of Difficult Mask Ventilation
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-101524-BO-ff
Record Dates: First submitted 2025-07-27; First posted 2025-08-11 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Airway Management; General Anesthesia; Mask Ventilation
Keywords: Airway management; Mask ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing general anaesthesia with facemask ventilation: Measurement of primary and secondary outcome parameters during induction of anaesthesia

SUMMARY:
The MASCAN Score is a prospectively developed objective classification for difficult facemask ventilation. This prospective observational study aims to externally validate the MASCAN score in patients undergoing general anaesthesia for surgical procedures and to determine the influence of different approaches and techniques, such as the timing of neuromuscular blocking agents and manual versus controlled facemask ventilation. A secondary aim is to determine the diagnostic value of visual assessments of the capnography curve. Another secondary aim of the study is to compare the assessment of the first attempt success during tracheal intubation between the airway operator and an independent observer.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for surgery with general anesthesia and require facemask ventilation and tracheal intubation after induction of anesthesia
* Patients aged 18 years or older
* Provided informed consent

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Required rapid sequence induction or other contraindications for facemask ventilation
* Planned awake tracheal intubation
* No consent given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive sampling: Adult patients undergoing general anesthesia in a tertiary care hospital who require facemask ventilation and tracheal intubation after induction of anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 926 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Difficult facemask ventilation | 1 hour
  Alert documented in patients health records by the airway operator following facemask ventilation

SECONDARY OUTCOMES:
Impossible facemask ventilation | 1 hour
  Impossible facemask ventilation observed after induction of anesthesia (absence of end-tidal carbon dioxide measurement and lack of perceptible chest wall movement despite airway adjuvants and additional personnel after adequate neuromuscular blockade)
Best capnograph achieved | 1 hour
  Best capnography waveform achieved during facemask ventilation (grade A-D)
Optimization manoeuvers for facemask ventilation used | 1 hour
  Optimization manouvers such as oral airway, jaw-thrust or two-handed grip used as documented facemask ventilation
Leak fraction | 1 hour
  Leak fraction (leak volume/ tidal volume) during facemask ventilation
Tidal volume | 1 hour
  Tidal volume during facemask ventilation (ml)
Senior anaesthetist taking over | 1 hour
  Senior anaesthetist taking over facemask ventilation as documented after facemask ventilation
Timing of neuromuscular blocking agent | 1 hour
  Observed during airway management (before/ after facemask ventilation)
Ventilation mode during facemask ventilation | 1 hour
  Manual or controlled ventilation applied by the airway operator
Change of ventilation mode during mask ventilation | 1 hour
  Observed during mask ventilation (to manual or controlled)
Difficult tracheal intubation | 1 hour
  Multiple tracheal intubation attempts documented after tracheal intubation
Difficult laryngoscopy | 1 hour
  Observed difficult laryngoscopy with restricted glottis view documented after tracheal intubation
First attempt success | 1 hour
  Successful tracheal intubation with only one attempt observed during tracheal intubation
Number of intubation attempts | 1 hour
  Observed during airway management
Number of laryngoscopy attempts | 1 hour
  Observed during airway management
Glottic view during laryngoscopy | 1 hour
  Grading of the best view obtained using landmarks (6-stages)
Percentage of glottis opening | 1 hour
  Grading of the best view obtained during laryngoscopy (%)
VIDiAC Score | 1 hour
  Classification of difficult (video-)laryngoscopic intubation (total score -1 to 5)
Failed primary intubation technique | 1 hour
  First-choice tracheal intubation technique unsuccessful
Lowest peripheral oxygen saturation | 1 hour
  Observed during airway management (%)
Drop of peripheral oxygen saturation during facemask ventilation | 1 hour
  Observed during facemask ventilation (%)
Airway-related adverse events | 1 hour
  Laryngospasm, bronchospasm, larynx trauma, airway trauma, soft tissue trauma, oral bleeding, edema, dental damage, corticosteroid application, accidental esophageal intubation, aspiration, hypotension or hypoxia
Post-intubation recommendation for an intubation method | 1 hour
  Recommendation issued by the airway operator after airway management for either awake tracheal intubation, camera-assisted intubation, direct laryngoscopy or other techniques
Anaesthesia alert card issued | 1 hour
  Anaesthesia alert card issued by the airway operator after airway management
  Anaesthesia alert card issued by the airway operator after airwaymanagement
Difficult tracheal intubation alert | 1 hour
  "Difficult tracheal intubation alert" issued by the airway operator after tracheal intubation in health records

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg, Germany